CLINICAL TRIAL: NCT00437775
Title: Angiotensin Converting Enzyme Inhibitors & Angiotensin Receptor Blocker in the Treatment of Type 2 Diabetic Patients Adverse Drug Effects and Drug Interactions- a Survey in an Internal Medicine Department.
Brief Title: ACEIs and ARBs Treatment in Diabetic Patients -Drug Interactions and Adverse Drug Effects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 167/06
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-01

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus type 2; ACE Inhibitors; ARBs; Adverse drug effect
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Proteinuria is an expression of diabetic nephropaty in type 1 and type 2 patients. Hypertenshion treatment and decreasing urine protein excretion, slow down renal deterioration. Treating diabetic ,hypertensive patients with Angiotensin Converting Enzyme inhibitors (ACEi), Angiotensin receptor blockers (ARBs)is common practice. The aim of our work is to examine 1.The prevalence of ACE and ARB treatment in diabetic patients with or without hypertension.2. Adverse drug reactions of ACEi and ARBs alone or in combination.

DETAILED DESCRIPTION:
The study group- men and women with diabetes mellitus type 2,who were hospitalized in the department of internal medicine in Assaf- Harofeh Medical Center.

During hospitalization, data regarding the clinical history,chronic diseases and drugs were collected from the medical files. Blood tests results were recorded during hospitalization .The patients were asked about adverse drug effects.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients admitted to department of Internal Medicine in Assaf Harofeh Medical Center

Exclusion Criteria:

* Type 1 diabetes mellitus

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2007-01; Study Completion 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Ahuva Golik, Assoc. Prof., Study Director — Sackler School of Medicine, Tel-Aviv University; Alina Alperovich, B.Pharm, Principal Investigator — Assaf-Harofeh Medical Center; Lila Akivison, MSc.Pharm, Study Chair — Assaf-Harofeh Medical Center; Sofia Berkovitch, MSc. Pharm, Study Chair — Assaf-Harofeh Medical Center; Gabby Elbaz, MD, Study Chair — Assaf- Hrofech Medical Senter
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

REFERENCES:
- [Result] Winkelmayer WC, Zhang Z, Shahinfar S, Cooper ME, Avorn J, Brenner BM. Efficacy and safety of angiotensin II receptor blockade in elderly patients with diabetes. Diabetes Care. 2006 Oct;29(10):2210-7. doi: 10.2337/dc06-0570. PMID 17003295
- [Result] Andros V, Egger A, Dua U. Blood pressure goal attainment according to JNC 7 guidelines and utilization of antihypertensive drug therapy in MCO patients with type 1 or type 2 diabetes. J Manag Care Pharm. 2006 May;12(4):303-9. doi: 10.18553/jmcp.2006.12.4.303. PMID 16792436
- [Result] Burnier M, Zanchi A. Blockade of the renin-angiotensin-aldosterone system: a key therapeutic strategy to reduce renal and cardiovascular events in patients with diabetes. J Hypertens. 2006 Jan;24(1):11-25. doi: 10.1097/01.hjh.0000191244.91314.9d. PMID 16331093